CLINICAL TRIAL: NCT06334224
Title: Effects of Twice Daily Blood Flow Restriction Training on Muscle Swelling, Markers of Exercise Induced Muscle Damage and Inflammation: A Randomised Control Trial
Brief Title: Acute Physiological Responses to Twice Daily Blood Flow Restriction Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Defence Medical Rehabilitation Centre, UK (Other Government)
Collaborators: University of Bath (Other)
Responsible Party: Principal Investigator, Peter Ladlow, Higher Scientific Officer and Chief Investigator, Defence Medical Rehabilitation Centre, UK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2242/MODREC/23
Record Dates: First submitted 2024-03-07; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Muscle Weakness; Muscle Damage
Keywords: resistance training; blood flow restriction; exercise induced muscle damage; muscle swelling; occlusion
MeSH Terms: conditions — Muscle Weakness; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Two arm randomised control trial
Masking Description: Due to the nature of the intervention, it is not possible to blind participants or outcome assessors to the treatment allocation. There is also no effective sham condition available. This is a common limitation within all blood flow restriction training research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-load resistance training (Active Comparator): Twice-daily low load resistance training for four days
  Interventions: Other: Low load resistance training
- Blood flow restriction training (Experimental): Twice-daily low load resistance training with blood flow restriction for four days
  Interventions: Device: Low load resistance training with blood flow restriction

INTERVENTIONS:
Device: Low load resistance training with blood flow restriction — The intervention involves placing a pneumatic tourniquet system over the proximal thigh. The cuff is inflated to 80% of limb occlusion pressure during lower limb strengthening exercises. These exercises include leg press and knee extensor exercises. Four sets (30,15,15,15 repetitions) performed at 20% of one repetition maximum.
  Arms: Blood flow restriction training
Other: Low load resistance training — Leg press and knee extensor exercises. Four sets (30,15,15,15 repetitions) performed at 20% of one repetition maximum.
  Arms: Low-load resistance training

SUMMARY:
The Academic Department of Military Rehabilitation (ADMR) is currently conducting a pan-defence, randomised control trial (RCT) investigating the utility of twice daily blood flow restriction training in UK military personnel with persistent knee pain (NCT05719922). Due to logistical confinements, this pan-defence RCT is confined to collecting outcome data pre and post-intervention. Therefore, the acute physiological mechanisms which underpin adaptation will remain unknown.

Consequently, ADMR is undertaking an additional, single centre RCT which will compare the acute physiological responses to low load resistance training with and without the addition of blood flow restriction. Specifically, this study will elucidate the effect of twice daily blood flow restriction training on measures of muscle swelling, muscle damage and inflammation. This data may aid in the optimisation of blood flow restriction exercise prescription within UK Defence Rehabilitation and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 55 years
* Must not have performed regular lower-limb resistance training for the last 6 months (participants must have performed < 1 lower-limb resistance training session per week over the previous 6 months)
* DMRC Staff member (civilian or service personnel)

Exclusion Criteria:

* Any medical contraindication related to BFR*.
* Any current lower-limb musculoskeletal injury
* Restricted range of movement. i.e. Chronically locked knee or fixed flexion deformity.
* Any physical impairment or co-morbidities (including cardio-vascular disease) precluding the safe participation in the intervention and/or assessment procedures
* Non-musculoskeletal or serious pathological condition (i.e. Inflammatory arthropathy, infection or tumour).
* Use of any medication which may contraindicate the performance of BFR or influence blood biomarkers of EIMD or inflammation.
* Use of any performance enhancing supplements or ergogenic aids such as creatine monohydrate.
* Any individual who is known to be currently pregnant

  *Medical-based Exclusion Criteria (based on clinical contraindications to performing BFR):
* History of cardiovascular disease (hypertension, peripheral vascular disease, thrombosis/embolism, ischaemic heart disease, myocardial infarction).
* History of the following musculoskeletal disorders: rheumatoid arthritis, avascular necrosis or osteonecrosis, severe osteoarthritis.
* History of the following neurological disorders: Peripheral neuropathy, Alzheimer's disease, amyotrophic lateral sclerosis, Parkinson's disease, severe traumatic brain injury.
* Varicose veins in the lower-limb.
* Acute viral or bacterial upper or lower respiratory infection at screening.
* Known or suspected lower limb chronic exertional compartment syndrome (tourniquet raises intra-compartmental muscle pressure).
* Postsurgical swelling.
* Surgical insertion of metal components at the position of cuff inflation.
* History of any of the following conditions or disorders not previously listed: diabetes, active cancer.
* History of elevated risk of unexplained fainting or dizzy spells during physical activity/exercise that causes loss of balance
* Increased risk of haemorrhagic stroke, exercise induced rhabdomyolysis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Maximum isometric voluntary contraction of knee extensor muscles | Measures collected in the morning on day 1,2,3,4,5,8. Measures also performed immediately before and 30 seconds after exercise on day 1 and 4
  Measured using an isokinetic dynamometer

SECONDARY OUTCOMES:
Vastus lateralis muscle thickness | Measures collected in the morning on day 1,2,3,4,5,8. Measures also performed before, 3 min after and 4 hours after exercise on day 1 and 4
  Measured using B-Mode ultrasound
Venous blood sampling for markers of exercise induced muscle damage | Measures collected in the morning on day 1,2,4,5,8. Measures also performed before, 10 min after and 4 hours after exercise on day 1
  Venous blood samples to measure markers of exercise induced muscle damage. E.g., Creatine Kinase (units/L)
Delayed onset muscle soreness | Measures collected in the morning on day 1,2,3,4,5,8
  Measured using a 100 mm visual analog scale. A higher score indicates greater levels of muscle soreness.
Quadriceps discomfort | Measured immediately after each exercise session
  Measured immediately after each exercise session using a 100 mm visual analog scale. A higher score indicates greater levels of discomfort.
Discomfort caused by the BFR cuff | Measured immediately after each exercise session
  Measured in the intervention group immediately after each exercise session using a 100 mm visual analog scale. A higher score indicates greater levels of discomfort.
Rating of perceived exertion | Measured immediately after each exercise session
  Measured using a Borg 0-10 rating of perceived exertion scale. A higher score represents greater levels of exertion.
Knee joint range of motion | Measures collected in the morning on day 1,2,3,4,5,8
  measured using a goniometer
Daily wellness questionnaire | Measures collected in the morning on day 1,2,3,4,5,8
  UK Defence Rehabilitation daily wellness questionnaire. This questionnaire asks participants to rate their: fatigue, muscle soreness, sleep quality, stress levels and mood on a 1-5 Likert scale.
Venous blood sampling for inflammatory markers | Measures collected in the morning on day 1,2,4,5,8. Measures also performed before, 10 min after and 4 hours after exercise on day 1
  Venous blood samples to measure markers of inflammation. E.g., Interleukin-6 (pg/ml), Tumour necrosis factor alpha (pg/mL) and vascular endothelial growth factor (pg/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bennett, PhD, Study Chair — Defence Medical Rehabilitation Centre
Locations (1):
- Defence Medical Rehabilitation Centre, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant data will be made available upon reasonable request to the chief investigator
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon completion of the dissemination of research findings (i.e., publications and conference proceedings)
Access Criteria: Most data will be openly available, but due to privacy concerns, some data regarding participants are available only to bona fide researchers working on a related project, subject to the completion of a non-disclosure agreement